CLINICAL TRIAL: NCT06419894
Title: Advanced Cardiac Magnetic Resonance Imaging for Assessment of Obstructive Coronary Artery Disease: ADVOCATE-CMR
Acronym: ADVOCATE-CMR
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Sonia Borodzicz-Jazdzyk, Project Leader, Amsterdam UMC, location VUmc
Other Study IDs: NL84828.015.23
Record Dates: First submitted 2024-05-03; First posted 2024-05-17 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: Stress perfusion cardiac magnetic resonance; Quantitative perfusion; Stress T1 mapping reactivity; Oxygen-sensitive cardiac magnetic resonance
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stress perfusion cardiovascular magnetic resonance (CMR) imaging is an established non-invasive imaging test for detection of obstructive coronary artery disease (CAD). Fully automated quantitative perfusion CMR (QP CMR) is a new technical advancement, which offers measurement of myocardial blood flow in CMR. Additionally, recent innovations have introduced various contrast-agent-free methods for CAD assessment, such as stress T1 mapping reactivity (∆T1) and oxygen-sensitive CMR (OS CMR). These methods might eliminate the necessity for contrast administration in clinical practice, simplifying, reducing time, invasiveness and costs in evaluating patients with suspected obstructive CAD. The ADVOCATE-CMR study aims to validate QP CMR, ∆T1 and OS CMR imaging against invasive fractional flow reserve (FFR) for detection of obstructive CAD. The study also aims to head-to-head compare the diagnostic accuracy of these CMR techniques with the conventional visual assessment of stress perfusion CMR and to correlate them to short- and long-term clinical outcomes.

DETAILED DESCRIPTION:
Study design: Single-center, observational, prospective, cross-sectional cohort study performed at the Amsterdam University Medical Centers - Location VUmc.

Study population: 182 symptomatic patients with suspected obstructive CAD (without a previous CAD history), scheduled for invasive coronary angiography (ICA) according to the decision of the treating clinician.

Methods:

1. CMR image acquisition prior to clinically scheduled ICA, using the following pulse sequences: cine imaging, OS-CMR with breathing maneuvers, adenosine-stress and rest T1 mapping, adenosine-stress and rest QP-CMR, late gadolinium enhancement;
2. Fractional flow reserve (FFR), instantaneous wave-free ratio (iFR), ratio between proximal and distal coronary pressures over entire resting cycle period (Pd/Pa ratio), coronary flow reserve (CFR) and index of microcircular resistance (IMR) in all main coronary arteries during ICA;
3. Follow-up CMR according to the abovementioned protocol 3 months after ICA (or 3 months after revascularization, if performed separately more than 1 day following ICA);
4. Clinical follow-up - 3, 6 months, 1 and 3 years after ICA or revascularization (if performed separately more than 1 day following ICA)

ELIGIBILITY:
Inclusion criteria:

* Suspected obstructive coronary artery disease
* No documented prior history of coronary artery disease
* Clinical referral for invasive coronary angiography according to the referring clinician's decision
* Competent adult (age ≥18 years)
* Signed informed consent

Exclusion criteria:

* Acute coronary syndrome
* History of coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting surgery)
* History of coronary artery disease or acute coronary syndrome (myocardial infarction, unstable angina)
* Use of sildenafil or dipyridamole that cannot be terminated
* Pregnancy or lactation
* Allergic reaction to iodized contrast
* Concurrent or prior (within last 30 days) participation in other research studies using interventional drugs
* Extensive comorbidities (i.e. cancer, other severe chronic diseases)
* Contraindication for cardiac magnetic resonance with gadolinium-based contrast agent (including severe claustrophobia, magnetic resonance unsafe implants/devices or MR conditional devices not suitable for 3T scanner, severe renal failure with estimated glomerular filtration rate<30 mL/min/1,73 m2, known hypersensitivity for gadolinium-based contrast agent)
* Contraindications for adenosine usage (including hypersensitivity to adenosine/dipyridamole/regadenoson, second or third degree atrio-ventricular block, sick sinus syndrome, sinus bradycardia (heart rate <40 bpm), long QT syndrome, severe hypertension (> 220/120 mmHg), systolic blood pressure <90mmHg, concomitant use of dipyridamole, severe asthma or severe chronic obstructive pulmonary disease)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 182 symptomatic patients with suspected obstructive CAD (without a previous CAD history), scheduled for invasive coronary angiography according to the decision of the treating clinician.
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2033-06-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of QP CMR (stress myocardial blood flow [MBF], stress relative MBF [rMBF], myocardial perfusion reserve [MPR] and relative MPR [rMPR]) to detect obstructive CAD, as defined by FFR | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, area under the curve (AUC), positive predictive value (PPV), negative predictive value (NPV)

SECONDARY OUTCOMES:
Diagnostic accuracy of ΔT1 to detect obstructive CAD, as defined by FFR | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Diagnostic accuracy of OS CMR (breathing-induced myocardial oxygenation reserve; B-MORE) to detect obstructive CAD, as defined by FFR | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Head-to-head comparison of diagnostic accuracies of QP CMR (stress MBF, stress rMBF, MPR, rMPR), ΔT1, OS CMR (B-MORE) and conventional visual assessment of GBCA-based first pass perfusion imaging to detect obstructive CAD, as defined by FFR | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Diagnostic accuracy of QP CMR (stress MBF, stress rMBF, MPR and rMPR) to detect obstructive CAD, as defined by iFR and resting Pd/Pa | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Diagnostic accuracy of ΔT1 to detect obstructive CAD, as defined by iFR and resting Pd/Pa | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Diagnostic accuracy of OS CMR (B-MORE) to detect obstructive CAD, as defined by iFR and resting Pd/Pa | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Head-to-head comparison of diagnostic accuracies of QP CMR (stress MBF, stress rMBF, MPR, rMPR), ΔT1, OS CMR (B-MORE) and conventional visual assessment of first pass perfusion imaging to detect obstructive CAD, as defined by iFR and resting Pd/Pa | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Relation of stress and rest MBF and rMBF, MPR and rMPR, ΔT1 and B-MORE to Seattle Angina Questionnaire (SAQ)-7 Summary score | Before ICA and 3, 6 months, 1 and 3 years after the ICA (or revascularization if applicable)
Relation of stress and rest MBF and rMBF, MPR and rMPR, ΔT1 and B-MORE to SAQ-7 Angina Frequency score | Before ICA and 3, 6 months, 1 and 3 years after the ICA (or revascularization if applicable)
Relation of stress and rest MBF and rMBF, MPR and rMPR, ΔT1 and B-MORE to SAQ-7 Physical Limitation score | Before ICA and 3, 6 months, 1 and 3 years after the ICA (or revascularization if applicable)
Relation of stress and rest MBF and rMBF, MPR and rMPR, ΔT1 and B-MORE to SAQ-7 Quality of Life score | Before ICA and 3, 6 months, 1 and 3 years after the ICA (or revascularization if applicable)
Relation of stress and rest MBF and rMBF, MPR and rMPR, ΔT1 and B-MORE to Rose Dyspnea Scale score | Before ICA and 3, 6 months, 1 and 3 years after the ICA (or revascularization if applicable)
Prognostic value of QP CMR (stress MBF, stress rMBF, MPR and rMPR), stress T1 mapping reactivity and OS CMR (B-MORE) | 3 months, 6 months, 1 year, 3 years
  1. Composite of cardiovascular (CV) death (death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, stroke, CV procedures, CV hemorrhage, other CV causes), myocardial infarction (according ESC/ACCF/AHA/WHF 4th Universal Definition of Myocardial Infarction), ischemia-driven coronary revascularization (all coronary revascularization performed in the context of myocardial infarction and those for worsening symptoms in combination with evidence of myocardial ischemia) or stroke (acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction);
  2. Composite of myocardial infarction or ischemia-driven coronary revascularization;
  3. Composite of cardiovascular death, stroke or myocardial infarction;
  4. Myocardial infarction;
  5. Ischemia-driven coronary revascularization;
  6. Stroke;
  7. Death from any cause;
  8. CV death

OTHER OUTCOMES:
Diagnostic accuracies of QP CMR (stress MBF, stress rMBF, MPR and rMPR), ΔT1 and B-MORE to detect microvascular dysfunction (MVD), as defined by CFR | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Diagnostic accuracy of QP CMR (stress MBF, stress rMBF, MPR and rMPR), ΔT1 and B-MORE to differentiate between MVD (as defined by CFR) and 3-vessel obstructive CAD | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Sensitivity, specificity, accuracy, AUC, PPV, NPV
Change in stress MBF after revascularization | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Difference between stress MBF before revascularization (baseline) and after revascularization (in ml/g/min)
Change in MPR after revascularization | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Difference between MPR before revascularization (baseline) and after revascularization
Change in stress T1 mapping after revascularization | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Difference between stress T1 mapping before revascularization (baseline) and after revascularization (in ms)
Change in ΔT1 after revascularization | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Difference between ΔT1 before revascularization (baseline) and after revascularization
Change in B-MORE after revascularization | ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
  Difference between B-MORE before revascularization (baseline) and after revascularization (in %)
Costs of QP CMR, stress T1 mapping reactivity and OS CMR compared to ICA | CMR and following ICA + hemodynamic measurements within 6 weeks of the initial CMR scan
Procedural time of QP CMR, stress T1 mapping reactivity and OS CMR compared to ICA | CMR and following ICA + hemodynamic measurements within 6 weeks of the initial CMR scan